CLINICAL TRIAL: NCT05093569
Title: Clinical Investigation of K'Watch - Lab & Home Study
Acronym: GLAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PKvitality (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT00014
Record Dates: First submitted 2021-09-29; First posted 2021-10-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Diabetes
Keywords: k'watch, diabetes,CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Iteration: 35 patients will be included in 7 iterations.
  Interventions: Device: K'watch

INTERVENTIONS:
Device: K'watch — Patients

SUMMARY:
This study categorized as a non significant risk trial is a monocentric, prospective, open-label comparative, paired-design trial aims to evaluate the performance and the tolerance of K'Watch CGM system in comparison with conventional reference (YSI system, BGM system and CGM systems ) . This trial will be conducted on patients with Type 1 and 2 of diabetes for 8 days.

DETAILED DESCRIPTION:
The purpose of this prospective study is to establish the performance and the cutaneous tolerance of the K'Watch device, for a Study Period of 8 hours (Lab-only study) to 8 days. This prospective study is divided in two phases: a first Laboratory phase will evaluate for 8 hours the safety and performance of the device under test (DUT) in a clinical controlled environment, then if no safety or critical performance issue occurred, the second phase will aim to collect data over a longer time frame, with the subjects using the DUT at home, and to get usability feedback for 6 additional consecutive days. This protocol is to evaluate a series of design iterations to K'Watch CGM system and its use on various populations.

All patients included will be followed for 28 days for safety requirements. 35 patients will be included in this trial and distributed in 7 iterations. For each iteration, the device tested will be improved according to the results obtained in the previous iteration.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male,
2. Subject with Type 1 Diabetes, or subject with Type 2 Diabetes (depending on the study iteration), - Type 1 Diabetes subjects taking insulin need to be on their current insulin regimen for ≥ 3 months prior to study entry,
3. Only patients using Dexcom device
4. Adult subjects, age 18 or older and ≤80 years,
5. Phototype: I to IV according to Fitzpatrick scale,
6. BMI ≤40 kg/m²,
7. Subject free from analgesics, anti-inflammatory drugs, antihistamines and/or local anesthetics within 7 days before inclusion and for the duration of the study,
8. Subject with a sufficient hand dexterity to apply the device,
9. Not practice vigorous physical exercise (running, fast cycling, aerobics) during the study period,
10. For subjects with Type 1 Diabetes, subjects must already be using a CGM (Abbott / Dexcom),
11. Willing to comply with the requirements of the study:

    * Self-administer Blood Glucose Measurements (BGM) in the frequency described in section 6.2.2 Blood Glucose Monitor (BGM),
    * Avoid swimming or taking a bath for the Study Period,
    * Use logbook to record adverse events and outcomes,
12. Wrist size in the range 16 - 21 cm,
13. Patients with hairiness grade between 1 to 3
14. Sufficient cooperation and understanding to comply with the study requirements,
15. Speak and read the English language,
16. Signed informed consent form prior to study entry.

Exclusion Criteria:

1. Subject with a known allergy to the components of the K'Watch CGM system (adhesive, disinfectants used during the study, ...),
2. Subject implanted with Active Medical device (Pacemaker, Defibrillator, any kind of active implantable medical devices that require active sensing to performed it intended use)
3. Subject suffering or having history of carpal tunnel syndrome,
4. Woman of childbearing potential not using an effective contraceptive, pregnant or breastfeeding,
5. Use of drugs that may interfere with glucose metabolism (such as steroids) unless they are chronic therapies whose dosage has remained stable over the past 3 months and is expected to remain stable during the study period,
6. Subject presenting, at the proposed application site, significant skin fragility/alterations/diseases that could interfere with the placement of the K'Watch CGM system. These conditions include, but are not limited to, history of skin irritation following the use of bandages or skin adhesives, extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scars, dermatitis herpetiformis, skin lesions, redness, infections or swelling,
7. Subject exercising a professional or a daily recreational activity involving immersion in the water of the K'Watch CGM system (e.g. lifeguard, plumber, …),
8. Subject with tattoos, piercings or implants at the proposed application site,
9. History of alcoholism (consumption of more than 5 "drinks" per day. For example, 12 ounces (35.5 cl) of beer, 5 ounces (15 cl) of wine, or 1 oz (4.5 cl) of distilled spirits,
10. Use of recreational drugs which would interfere with participation in the study, as determined by the PI,
11. Hair removal or shaving in the area of application of the K'Watch CGM system over the month prior to inclusion and throughout the duration of the study,
12. Application of cosmetics on the application area of the device the day before the Lab phase and during the Study Period,
13. Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen during the study,
14. Subject with a scheduled radiographic, MRI, CT or diathermy appointment during the study participation period, and the appointment cannot be postponed,
15. Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or clinical staff,
16. Subject currently is participating in another clinical trial,
17. European citizen. (PK will not recruit european citizens for this trial, because the sponsor prefer not to implement the additional administrative steps as required by the GDPR).
18. Prisoners or subjects who are involuntarily incarcerated

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Type 1 and 2 of diabetes
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
to determine the accuracy of K'Watch Release 0.x CGM system glucose readings at day 1 as compared to standard references. | 14 months
  The Primary endpoint in this trial is the degree of compliance with the accuracy section of the FDA Class II Integrated continuous glucose monitoring (iCGM) requirements after one entire day.

SECONDARY OUTCOMES:
Accuracy of the investigational device compared to the standard reference CGM devices | Between day1 and day 7
  Accuracy of the investigational device compared to the standard reference CGM devices by measuring the median absolute relative difference (MARD)
The number and duration of gaps in sensor data availability | 14 months
  This is intended to measure the time that the sensor was not able to measure glucose, even though the watch was connected. If the user removes the watch, then this time is not considered to be a "gap"
Safety of the K'Watch system, characterizing device-related Adverse Events | 14 months
  Safety of the K'Watch system, characterizing device-related Adverse Events
Safety of the K'Watch system characterizing device-related pain intensity (Visual Analogue Scale scores from 0-10) recorded during the study. | 14 months
  Safety of the K'Watch system characterizing device-related pain intensity (Visual Analogue Scale scores from 0-10) recorded during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- AMCR Institute, San Diego, California, United States